CLINICAL TRIAL: NCT05021614
Title: Evaluation of the Efficacy and Safety of the Transcatheter Mitral Valve Repair System in Patients With Moderate and Above Degenerative Mitral Regurgitation at High Surgical Risk
Brief Title: Valveclip® Transcatheter Mitral Valve Repair Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai NewMed Medical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M-clip-2020-09
Record Dates: First submitted 2021-08-16; First posted 2021-08-25 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Mitral Regurgitation
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Transcatheter Mitral Valve Repair with Valveclip®
  Interventions: Device: Valveclip® Transcatheter mitral valve repair

INTERVENTIONS:
Device: Valveclip® Transcatheter mitral valve repair — Transcatheter mitral valve repair system

SUMMARY:
The purpose of this clinical trial is to evaluate the effectiveness and safety of the transcatheter mitral valve repair system in the treatment of patients with moderate or above degenerative mitral regurgitation.

DETAILED DESCRIPTION:
This study is a prospective,multi-center, single-arm, safety and performance clinical study.

ELIGIBILITY:
Inclusion Criteria:

1. Severe mitral regurgitation≥3+ (moderate or above degenerative mitral regurgitation disease, or with stenosis is included);
2. Age≥70 years; or patients who are 60~70 years old, and the STS risk score indicate that participants are at high risk of traditional surgery or cannot tolerate traditional thoracotomy;

4) Left ventricular ejection fraction≥30%； 5) As assessed by multidisciplinary cardiac team (at least two cardiac surgeons/one cardiologist), patients who are at extremely high-risk or unsuitable for routine mitral valve surgery with evaluation; 6) Patients who understand the purpose of the trial and volunteer to participate in, sign the informed consent form and are willing to accept relevant examinations and clinical follow-ups.

Anatomy selection Criteria：

1. The regurgitant jet of mitral valve originates from the A2 and P2 (the lesions of A2/P2 in mitral valve causes regurgitation);
2. The width of the mitral valve prolapsed area is ≤15mm, Height of Prolapse ≤10mm or coaptation depth≤11mm, coaptation height≥2mm, effective length of anterior and posterior leaflets>1cm (conforming to EVEREST II recommended mitral valve interventional edge-to-edge repair standards);
3. Effective mitral valve orifice area≥ 4.0cm2;
4. No obvious calcification of the mitral valve annulus and valve leaflets;
5. Patient's anatomical conditions allow transseptal approach.

Exclusion Criteria:

1. Previous cardiac mitral valve surgery;
2. Patients with Infective endocarditis or having an active infection;
3. Patients with mitral regurgitation caused by pure mitral stenosis;
4. Combined with untreated severe coronary artery disease
5. Pulmonary hypertension (pulmonary artery systolic pressure>70mmHg);
6. Patients with severe right heart failure;
7. Patients are extremely weak and cannot tolerate general anesthesia or are in shock that circulatory support is needed;
8. Patients with hypertrophic cardiomyopathy, restrictive cardiomyopathy, and constrictive pericarditis;
9. Patients receiving chronic dialysis;
10. Patients with clear coagulation dysfunction and severe coagulopathy;
11. Patients with clear contraindications to anticoagulant drugs;
12. Patients with stroke or transient ischemic attack within 30 days;
13. Echocardiography found any intracardiac mass, left ventricle or atrial thrombus;
14. Patients who require surgery or interventional therapy for other valvular lesions;
15. Patients with severe macrovascular lesions requiring surgical treatment;
16. Patients' imaging examinations suggest that the anatomy of the heart and valves are inappropriate;

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-09-24 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Efficacy of product | 12 months
  Efficacy of product is defined as the proportion of participants meeting effective standards after surgery (freedom from death, mitral valve reoperation or MR>2+ at 12 months).

SECONDARY OUTCOMES:
Efficacy of product | 30 days, 180 days, 2 to 5 years
  Efficacy of product is defined as the proportion of participants meeting effective standards after surgery (freedom from death, mitral valve reoperation or MR>2+ at 30 days, 180 days, 2 to 5 years).
Rate of Cardiovascular related mortality | 30 days, 180 days, 1 year, 2 to 5 years
  Cardiovascular related mortality after Transcatheter Mitral Valve Repairment
Rate of Severe adverse events | 30 days, 180 days, 1 year, 2 to 5 years
  Severe adverse events after Transcatheter Mitral Valve Repairment (including death, stroke, myocardial infarction, reoperation, instrumental non-selective cardiovascular surgery, renal failure, and adverse events related to transfemoral vein septal approach surgery, etc.）
Quality of life Improvement | 30 days, 180 days, 1 year, 2 to 5 years
  The 12-Item Short-Form Health Survey(SF-12)

OTHER OUTCOMES:
Technical success | immediate post-surgical
  Technical success after Transcatheter Mitral Valve Repairment
Device success | 30 days、180 days、1 year
  Device success after Transcatheter Mitral Valve Repairment
Procedural success | 30 days
  Procedural success after Transcatheter Mitral Valve Repairment

CONTACTS AND LOCATIONS:
Overall Officials: mao Chen, Chief, Principal Investigator — West China Hospital
Locations (1):
- Department of Cardiology, West China Hospital, Sichuan University, Sichuan, China

IPD SHARING:
Plan to Share IPD: No